CLINICAL TRIAL: NCT01124760
Title: A Phase I, Single Center, Open Label, 2-consecutive-group, 2-period, 1-sequence Crossover Study to Assess the Effect of Diltiazem (Cardizem), a Moderate CYP3A4 Inhibitor, or Ketoconazole, a Potent CYP3A4 Inhibitor, on the Pharmacokinetics of a Single Intravenous Dose of 150mg of AZD9742.
Brief Title: Open Label Study, Assessing the Effect of Diltiazem or Ketoconazole on the Pharmacokinetics of AZD9742 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D2690C00008
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Pharmacokinetics
Keywords: open label; 2-consecutive-group; 2-period; 1-sequence crossover study
MeSH Terms: interventions — Diltiazem; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): AZD9742
  Interventions: Drug: AZD9742; Drug: Diltiazem; Drug: ketoconazole

INTERVENTIONS:
Drug: AZD9742 — Sterile solution, 620 mg (20 mg/mL) in 50 mL vial with a fill volume of 31 mL; On Day 7, a single 150 mg IV dose, coadministered after the morning dose of ketoconazole
Drug: Diltiazem — Orally, daily beginning on Day 4 for 14 consecutive days
  Other Names: Myoderm
Drug: ketoconazole — 200 mg, orally, every 12 hours starting on Day 4 for 10 consecutive days in which on Day 13 only the morning dose will be administered

SUMMARY:
The aim of this study is to examine the effect of coadministration of CYP3A4 inhibitors on the pharmacokinetics of AZD9742.

ELIGIBILITY:
Inclusion Criteria:

* non-childbearing potential, with suitable veins for cannulation or repeated venipuncture
* Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening.
* Male volunteers should be willing to use barrier contraception, ie, condoms, from the day of dosing until 3 months after dosing with the investigational product.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs as judged by Investigator.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational product

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the effect of coadministration of CYP3A4 inhibitors (diltiazem and ketoconazole) on the pharmacokinetics of AZD9742 in blood and urine. | For diltiazem group - up to 18 days of pre-defined study days for pk profiling. For keoconazole - up to 14 days of pre-defined study days for pk profiling.

SECONDARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examinations, clinical laboratory assessments, 12-lead ECG, telemetry) | Collected prior to treatment, during treatment, and follow-up for a maximum of 57 days for group 1 and 53 days for group 2 (this includes up to 28 days for screening).

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Schutz, MD, Principal Investigator — Quintiles, Inc.; Colleen Jensen, Study Director — AstraZeneca; Brendan Smyth, Study Chair — AstraZeneca
Locations (1):
- Research Site, Overland Park, Kansas, United States